CLINICAL TRIAL: NCT02848079
Title: TAS-102 and Oxaliplatin (TAS-OX) for Refractory Metastatic Colon Cancer
Brief Title: TAS-OX for Refractory Metastatic Colon Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1605017852
Record Dates: First submitted 2016-07-21; First posted 2016-07-28 (Estimated); Results first posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- combined TAS-102 and oxaliplatin (Experimental): Combination treatment with TAS-102 and oxaliplatin. Combination treatment with TAS-102 and oxaliplatin. TAS-102 is an oral medication; oxaliplatin (TAS-OX) is given by infusion. In Part 1 treatments were started at level 1 doses, which were based on prior clinical experience with the medications studied. Dose escalation followed a traditional "3+3" design. The subjects in Part 2 were treated with dose level 3.
  Oxaliplatin infusion was given on day 1 of each cycle. TAS-102 was taken twice daily on days 1-5 of each cycle.
  Interventions: Drug: combined TAS-102 and TAS-OX

INTERVENTIONS:
Drug: combined TAS-102 and TAS-OX — Combination treatment with TAS-102 and oxaliplatin. TAS-102 is an oral medication; oxaliplatin (TAS-OX) is given by infusion.

SUMMARY:
This study will examine the safety and effectiveness of oxaliplatin in combination with TAS-102 (TAS-OX) for treatment of patients with metastatic colorectal cancer whose cancer has progressed or recurred after FOLFOX chemotherapy.

DETAILED DESCRIPTION:
TAS-102 is an oral agent, which consists of a combination of a novel antimetabolite 5-trifluorothymidine (FTD) and a thymidine phosphorylase inhibitor (TPI) that prevents degradation of FTD. It has demonstrated activity in chemorefractory metastatic colorectal cancer (mCRC) patients. In the Japanese randomized phase II trial, TAS-102 improved medial overall survival when compared to placebo (9.0 vs.6.6 months, Hazard Ratio (HR) 0.56) in patients with mCRC refractory to 5-fluorouracil (5-FU), irinotecan and oxaliplatin. Subsequently, a randomized phase III study conducted in 13 countries (RECOURSE trial) confirmed this benefit on overall survival when compared to placebo (7.1 months vs. 5.3 months, HR 0.68) in patients with refractory metastatic colorectal cancer (CRC) 5.

Oxaliplatin is a third generation platinum compound, which is active when used together with 5-FU in the treatment of mCRC (FOLFOX). FOLFOX chemotherapy, which is frequently combined with anti-angiogenic agent Bevacizumab, is widely accepted as the preferred first-line regimen in the treatment of this disease in the US. Oxaliplatin is also frequently reintroduced in more advanced settings. Reintroduction is seen after progression on maintenance therapy, after resolution of previous treatment limiting neuropathy, after disease recurrence post adjuvant treatment or post metastasectomy. In the control arm of a randomized study of FOLFOX4 or FOLFOX7 with oxaliplatin in a stop-and-go fashion in advanced colorectal cancer (OPTIMOX1 study), oxaliplatin was reintroduced in 27% of patients. Although patients derive clinical benefit when oxaliplatin is reintroduced, the response rates are not as robust as during initial exposures. Decreased efficacy may be at least in part due to prolonged exposure and resultant resistance to 5-FU, which is a backbone in maintenance and in oxaliplatin containing regimens. Hence, the investigators propose exploring the safety and efficacy of oxaliplatin in combination with an alternative anti-metabolite TAS-102 (TAS-OX).

TAS-102 has demonstrated activity in 5-FU refractory mCRC, so the investigators hypothesize that TAS-OX may serve as an alternative drug combination for patients who have progressed or recurred after FOLFOX, and who are candidates for additional oxaliplatin therapy.

This is a 2-part clinical trial with TAS-102 in combination with oxaliplatin. The first part will be a dose-finding run-in phase and will enroll 3-18 patients. The second part, the focus of this study, will be a single arm cohort , which will further evaluate the safety, as well as efficacy, of TAS-OX in the treatment of mCRC. The subjects in part 2 will be treated with the drug doses determined in Part 1 of the trial. Up to 50 patients will be enrolled in part 2. Anticipated enrollment may be as high as 68 patients. Maximum potential enrollment is listed under anticipated enrollment, below.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed stage IV colon cancer (AJCC 7th edition) that has progressed after standard therapy that included 5-FU, irinotecan and oxaliplatin. Patients who could not tolerate standard agents because of unacceptable, but reversible, toxicity necessitating their discontinuation will be allowed to participate.
2. Patients who had received adjuvant chemotherapy and had recurrence during or within 6 months of completion of the adjuvant chemotherapy will be allowed to count the adjuvant therapy as one chemotherapy regimen.
3. Progression of disease must be documented on the most recent scan.
4. Presence of measurable disease (not required for Phase 1 portion of the trial).
5. Retrovirus-associated DNA sequences (RAS) mutation and mismatch repair (MMR) status must be determined (or tissue availability for testing if not already determined)
6. Age 18 years or older.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
8. Life expectancy of at least 3 months.
9. Patient with adequate organ function:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   2. Hemoglobin ≥ 9 g/dL
   3. Platelets (PLT) ≥ 75 x 109/L
   4. Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) ≤ 5 x Upper limit of normal (ULN)
   5. Total serum bilirubin of ≤1.5 mg/dL (except for Grade 1 hyperbilirubinemia due solely to a medical diagnosis of Gilbert's syndrome).
   6. Albumin ≥ 2.5 g/dL
   7. Serum creatinine ≤ 1.5 x institutional ULN (Cockcroft and Gault formula)
10. Adequate contraception if applicable.
11. Women who are nursing must discontinue nursing prior to enrollment in the program.
12. Ability to take oral medication (i.e. no feeding tube).
13. Patient able and willing to comply with study procedures as per protocol.
14. Patient able to understand and willing to sign and date the written voluntary informed consent form (ICF) at screening visit prior to any protocol-specific procedures.

Exclusion Criteria:

1. Patients who have previously received TAS-102.
2. Grade 2 or higher peripheral neuropathy.
3. Symptomatic Central nervous system (CNS) metastases requiring treatment.
4. Other active malignancy within the last 3 years (except for non-melanoma skin cancer or a non-invasive/in situ cancer).
5. Pregnancy or breast feeding.
6. Current therapy with other investigational agents.
7. Active infection with body temperature ≥38°C due to infection.
8. Major surgery within prior 4 weeks (the surgical incision should be fully healed prior to drug administration).
9. Any anticancer therapy within prior 3 weeks of first dose of study drug.
10. History of allergic reactions attributed to compounds of similar chemical or biologic composition to TAS-102.
11. Current therapy with other investigational agents or participation in another clinical study or any investigational agent received within prior 4 weeks.
12. Grade 3 or higher hypersensitivity reaction to oxaliplatin, or grade 1-2 hypersensitivity reaction to oxaliplatin not controlled with pre-medication.
13. Unresolved toxicity of greater than or equal to Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 attributed to any prior therapies (excluding anemia, alopecia, skin pigmentation, and platinum-induced neurotoxicity).
14. Extended field radiation within prior 4 weeks of first dose of study drug or limited field radiation within prior 2 weeks of first dose of study drug.
15. Psychological, familial, or sociological condition potentially hampering compliance with the study protocol and follow-up schedule.
16. Involvement in the planning and/or conduct of the study.
17. Previous enrollment in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy S. Kortansky, M.D., Principal Investigator — Yale University
Locations (1):
- Yale Cancer Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined TAS-102 and TAS-OX: Combination treatment with TAS-102 and oxaliplatin. TAS-102 is an oral medication; oxaliplatin (TAS-OX) is given by infusion. In Part 1 treatments were started at level 1 doses, which were based on prior clinical experience with the medications studied. Dose escalation followed a traditional "3+3" design. The subjects in Part 2 were treated with dose level 3.
  Oxaliplatin infusion was given on day 1 of each cycle. TAS-102 was taken twice daily on days 1-5 of each cycle.
Period: Overall Study
Arm/Group | Combined TAS-102 and TAS-OX
Started | 41
Receieved Study Treatment | 41
Discontinued | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Combined TAS-102 and TAS-OX
Number analyzed (Participants) | 41
Age, Customized [Median (Full Range); unit: years] | 62 [42 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 38
  Black | 1
  Asian | 2
ECOG [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status is used to determine performance status.
  A score of "0" is defined as - Fully active, able to carry on all pre-disease performance without restriction A score of "1" is defined as - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work.
  Participants
    0 | 25
    1 | 16
Location of primary tumor, No. [Count of Participants; unit: Participants]
  Left side of colon, including rectum | 31
  Right side of colon | 10
Stage at diagnosis [Count of Participants; unit: Participants] — Stage at diagnosis was assessed using AJCC version 7. The lower the number, the less the cancer has spread.
  Participants
    I | 1
    II | 2
    III | 13
    IV | 25
Histology [Count of Participants; unit: Participants]
  Well-differentiated | 2
  Moderately differentiated | 30
  Poorly differentiated | 9
High microsatellite instability [Count of Participants; unit: Participants] | 2
KRAS/BRAF mutation [Count of Participants; unit: Participants]
  KRAS mutation | 20
  BRAF mutation | 1
  Wild type | 20
Number of prior therapies [Count of Participants; unit: Participants] — The number of prior therapies a patient had received at baseline assessment.
  Participants
    1 therapy | 1
    2 therapies | 18
    3 therapies | 15
    ≥ 4 therapies | 7
Progression during prior oxaliplatin [Count of Participants; unit: Participants]
  Yes | 18
  No | 23

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall Response Rate was measured by Response Evaluation Criteria In Solid Tumor (RECIST) 1.1 criteria. Tumors were assessed with CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.".
Time Frame: up to 30 days following discontinuation of treatment
Population: Intention-to-treat (ITT)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combined TAS-102 and TAS-OX
Number analyzed (Participants) | 41
months | 2.4 [0 to 12.9]

2. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival was assessed according to RECIST criteria version 1.1. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: from the date of start of treatment to the date of first documented progression or any cause of death assessed up to 12 months.
Population: Intention-to-treat (ITT)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combined TAS-102 and TAS-OX
Number analyzed (Participants) | 41
months | 2.7 [2.4 to 4.8]

3. Secondary Outcome: Overall Survival
Description: Overall Survival was assessed by the time to death from start of study.
Time Frame: from the date of start of treatment to the date of any cause of death assessed up to 24 months.
Population: Intention-to-Treat (ITT)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combined TAS-102 and TAS-OX
Number analyzed (Participants) | 41
months | 6.8 [5.4 to 10.0]

ADVERSE EVENTS:
Time Frame: up to 38 months
Description: The reported AEs here are all AEs in the study, regardless of attribution. Whereas in the published manuscript, SAE's were reported when they could be attributed to treatment and that a 10% threshold was used in reporting AE's.
Arm/Group | Combined TAS-102 and TAS-OX
All-Cause Mortality (participants affected / at risk) | 37/41
Serious Adverse Events (participants affected / at risk) | 8/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combined TAS-102 and TAS-OX (N=41)
Fever (General disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Failure to thrive
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 — Intrahepatic biliary ductal dilation
Infections and infestations - Other, specify (Infections and infestations) | 1 — Perirectal abcess
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 — Hydroureteronephrosis
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 — Post-influenza pneumonia
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined TAS-102 and TAS-OX (N=41)
Diarrhea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 12 (20)
Peripheral sensory neuropathy (Nervous system disorders) | 6
Anorexia (General disorders) | 16 (21)
Anemia (Blood and lymphatic system disorders) | 25 (46)
Neutrophil count decrease (Investigations) | 15 (49)
Platelet count decrease (Blood and lymphatic system disorders) | 13
White blood cell decreased (Investigations) | 14 (51)
Alkaline phosphatase increased (Blood and lymphatic system disorders) | 20 (28)
Abdominal Pain (Gastrointestinal disorders) | 11 (14)
Alanine aminotransferase increased (Investigations) | 9 (12)
Aspartate aminotransferase increased (Investigations) | 14 (22)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 8 (24)
Blood bilirubin increased (Investigations) | 10 (22)
Constipation (Gastrointestinal disorders) | 11 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (12)
Creatinine increased (Investigations) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 13 (24)
Dizziness (Nervous system disorders) | 6 (7)
Dysgeusia (Nervous system disorders) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Fatigue (General disorders) | 27 (48)
Fever (General disorders) | 4 (6)
Flatulence (Gastrointestinal disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Hypertension (Vascular disorders) | 12 (23)
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 (17)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (8)
Hypokalemia (Metabolism and nutrition disorders) | 7 (9)
Hyponatremia (Metabolism and nutrition disorders) | 12 (17)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (7)
INR increased (Investigations) | 4 (11)
Insomnia (Psychiatric disorders) | 7 (9)
Lymphocyte count decreased (Investigations) | 15 (49)
Nausea (Gastrointestinal disorders) | 22 (39)
Pain (General disorders) | 3 (5)
Paresthesia (Nervous system disorders) | 8 (13)
Peripheral sensory neuropathy (Nervous system disorders) | 17 (24)
Platelet count decreased (Investigations) | 17 (59)
Sinusitis (Infections and infestations) | 3 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (3)
Weight Loss (Investigations) | 4 (5)
Edema limbs (General disorders) | 6 (8)
Infusion related reaction (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT02848079/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT02848079/ICF_001.pdf